CLINICAL TRIAL: NCT04675541
Title: Observational Register of Patients With haEmophilia A tReated With Afstyla®
Brief Title: Register of Patients With haEmophilia A tReated With Afstyla®
Acronym: OPERA
Status: Completed | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: OPERA study; 2017-A03517-46 (Other: ANSM)
Record Dates: First submitted 2020-12-01; First posted 2020-12-19 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Haemophilia A
Keywords: FVIII; Coagulation FVIII
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Afstyla® — Solution for injection
  Other Names: CSL627

SUMMARY:
Record real life data of patients with Hemophilia A and treated with Afstyla® to assess the effectiveness and the safety of the treatment used as prophylaxis, prevention of bleeding (e.g. surgery) or on-demand treatment during 3 years after patient inclusion

DETAILED DESCRIPTION:
Haemophilia A is a congenital coagulation disorder caused by a deficiency or abnormality of coagulation factor VIII (FVIII).

The severity of the haemophilia depends on the magnitude of the FVIII deficiency and the clinical features depend on the site of the bleed.

The therapeutic management of this disease involves administering the deficient factor, FVIII to the patient. Depending on the severity of the disease and patient background, the management regimens are different (long term prophylactic treatment to prevent non surgical bleeds, prophylactic short term treatment to prevent surgical bleeds or treatment of acute bleeds on demand).

Several recombinant or plasma derived treatments are currently available. The CSL Behring Company has designed a new recombinant single chain B1FVIII, rFVIII (Afstyla®). This has increased affinity for VWF, resulting in improved stability and an improvement in its pharmacokinetic indices. OPERA is a non-interventional, prospective and national study which aim is to record real life data in haemophilia A French patients treated with Afstyla® in order to confirm the efficacy and safety of this proprietary product established in clinical development studies.

ELIGIBILITY:
Inclusion Criteria:

* Have given their agreement to take part in the observational registry after being informed in writing of the purposes of the study and after their data have been recorded (parent's agreement for minor patients);
* Be suffering from haemophilia A and being treated or having been treated with Afstyla® long term prophylactically, on demand or preventatively for a surgical procedure;
* Absence of inhibitor and/or treatment for immune tolerance at the time of inclusion

Exclusion Criteria:

* Refusal of the patient or the patient's legal representative to take part in the study;
* Existence of a contraindication to the use of Afstyla® treatment (known hypersensitivity to FVIII or hamster proteins);
* Simultaneous participation in an interventional clinical study.
* Presence of an inhibitor and/or ongoing immune tolerance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Haemophilia A French patients treated with Afstyla®
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The annualized bleeding rate (spontaneous, traumatic) during long term prophylactic and on demand regimen. | Up to 36 months
The number of spontaneous bleeding episodes per patient | Up to 36 months
The number of infusions of Afstyla® required for the prevention and resolution of non-surgical bleeding episodes | Up to 36 months
The total dose of Afstyla® required for the prevention and resolution of non-surgical bleeding episodes | Up to 36 months

SECONDARY OUTCOMES:
The number of infusions of Afstyla® required during the surgical procedures | Up to 36 months
The total dose of Afstyla® required during the surgical procedures | Up to 36 months
The incidence of adverse events (AE), severe AE, and AE related to Afstyla® | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring SA
Locations (17):
- France (17):
  - CHU Brest, Brest
  - CHU Caen, Caen
  - CHU Chambéry, Chambéry
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Simone Veil, Eaubonne
  - Hôpital Mignot, Le Chesnay
  - CRC-MHC Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Hôpital Necker, Paris
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU Saint-Etienne, Saint-Etienne
  - Hôpital Hautepierre, Strasbourg
  - CHRU de Tours, Tours